CLINICAL TRIAL: NCT01306006
Title: The Effect on Overall Mortality of a National Policy of Limiting Measles Vaccination to Children Below 12 Months of Age
Acronym: MVEPI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Institudo Nacional de Saude Publica INASA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MV-EPI
Record Dates: First submitted 2011-02-24; First posted 2011-03-01 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mortality; Vaccines
Keywords: Mortality; Vaccines

ARMS (2):
- MV-for-all (Active Comparator): Measles vaccine provided to all children aged 9 months -3 years of age
  Interventions: Biological: Providing measles vaccine for all children 9-35 months who have not yet received a routine measles vaccine
- National policy (No Intervention): Measles vaccine provided to children aged 9-11 months, if there are sufficient children to open a measles vaccine vial.

INTERVENTIONS:
Biological: Providing measles vaccine for all children 9-35 months who have not yet received a routine measles vaccine — Normal measles vaccines licensed for distribution through the national EPI program
  Arms: MV-for-all

SUMMARY:
The national Expanded Programme on Immunization (EPI) in Guinea-Bissau focuses its efforts exclusively on children below 12 months of age; children who have reached 12 months of age are no longer entitled to vaccines through the EPI program. This has affected the measles vaccination coverage, approx. 30% of the children in the rural area do not receive measles vaccine (MV).

Studies from the Bandim Health Project (BHP) have shown that MV has a profound impact on survival, reducing mortality by approximately 50% - far more than can be explained by prevention of measles deaths. Hence, MV seems to have non-specific beneficial effects on survival, and the current policy may have important consequences for overall child mortality.

To test the implications of the current policy of only vaccinating children below 12 months of age, the investigators will conduct a cluster randomized trial, in which children will receive their vaccines according to the current national EPI policy (National policy) or receive MV regardless of age and whether some doses of MV may be lost (MV-for-all policy).

The investigators hypothesise that among children enrolled after 12 months of age, mortality is 50% lower in children randomised to receive MV compared with children randomised to follow the national policy and not receive MV.

ELIGIBILITY:
Inclusion Criteria:

* Age 9-35 months, not yet received routine measles vaccination, resident in study area

Exclusion Criteria:

* To ill to be vaccinated (according to local practice)

Ages: 9 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3500 (Estimated)
Dates: Start 2011-02 (Actual); Primary Completion 2017-12-02 (Actual); Study Completion 2017-12-02 (Actual)

PRIMARY OUTCOMES:
Mortality

SECONDARY OUTCOMES:
Hospital morbidity

CONTACTS AND LOCATIONS:
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

REFERENCES:
- [Result] McClure BA, Du H, Liu YH, Clarke AE. S-locus products in Nicotiana alata pistils are subject to organ-specific post-transcriptional processing but not post-translational processing. Plant Mol Biol. 1993 Apr;22(1):177-81. doi: 10.1007/BF00039008. PMID 8098964
- [Derived] Byberg S, Aaby P, Rodrigues A, Stabell Benn C, Fisker AB. The mortality effects of disregarding the strategy to save doses of measles vaccine: a cluster-randomised trial in Guinea-Bissau. BMJ Glob Health. 2021 May;6(5):e004328. doi: 10.1136/bmjgh-2020-004328. PMID 33941513
- See also: Related Info — http://www.bandim.org